CLINICAL TRIAL: NCT06510179
Title: Effectiveness of Different Types of Toothbrushes on Periodontal Health in Orthodontic Patients With Gingivitis: a Randomized Controlled Study
Brief Title: Effectiveness of Different Types of Toothbrushes on Periodontal Health in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, GOKCE AYKOL SAHIN, Assistant professor, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/30 Rev-1/ 681
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Gingivitis; Orthodontics
Keywords: orthodontic appliances; oral hygiene; toothbrushing; gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Toothbrushing

STUDY DESIGN:
Intervention Model Description: Patients will randomly allocate one of three groups (Conventional toothbrush group, orthodontic toothbrush group, or single-tufted toothbrush group).
Who Masked: Investigator
Masking Description: The researcher performing the clinical examination will not know the group in which the patients are included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional toothbrush group (Active Comparator): Patients are instructed with the modified Bass technique. In this technique, the toothbrush bristles are positioned 45° to the long axis of the tooth towards the base of the tooth at the gum line with a gentle back-and-forth rolling motion, then swept towards the occlusal surface of the teeth. To adapt to orthodontic braces, the same movement is repeated with the bristles positioned just occlusal to the brackets.
  Interventions: Other: Toothbrushing
- Orthodontic toothbrush group (Experimental): The patients in this group are instructed to brush with the Bass technique. In this technique, the toothbrush is placed on the gingival margin with its bristles at 45° to the long axis of the tooth. It is demonstrated by making back-and-forth movements and vibrating the brush at short intervals without lifting the bristles.
  Interventions: Other: Toothbrushing
- Single-tufted toothbrush group (Experimental): In this group, a single-tooth circular brushing technique first developed by Jiri Sedelmayer was explained, and dental plaque removal is demonstrated with circular movements around the brackets and following the gingival margin of each tooth.
  Interventions: Other: Toothbrushing

INTERVENTIONS:
Other: Toothbrushing — Patients brush their teeth using the technique instructed to them using the toothbrush provided.

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of different toothbrushes in patients with fixed orthodontic appliances who have gingival inflammation. The main questions it aims to answer are:

1. Is a single-tufted toothbrush as effective as orthodontic or conventional toothbrushes?
2. What are the effects of these toothbrushes on dental biofilm removal and gingival inflammation? Researchers will compare conventional toothbrushes, orthodontic toothbrushes, and single-tufted toothbrushes after professional mechanical debridement and oral hygiene instruction.

Participants will:

1. Receive nonsurgical periodontal therapy
2. According to the group they are involved, they will receive an oral hygiene kit (toothbrush and toothpaste) and instruction
3. They will participate in the recalls in the first week, sixth week, and third month.

DETAILED DESCRIPTION:
Fixed orthodontic treatment is often the preferred method for the treatment of malocclusion and involves using complex devices like brackets and arch wires. These devices create areas that retain plaque, making effective plaque removal more challenging. Studies have shown that patients with fixed orthodontic appliances tend to have increased plaque accumulation.1,2 These patients are more susceptible to gingival inflammation due to this plaque-accumulating environment. The essential role of dental biofilm in gingivitis is well-documented, and removing biofilm can reverse the condition.3 Previous animal studies on dentition with reduced periodontium have shown that orthodontic forces and tooth movements do not induce gingival inflammation without plaque.4-7 However, in the presence of plaque, similar forces can result in vertical bone defects and attachment loss, especially with tipping and intruding movements.4 Effective dental biofilm control is crucial for improving oral hygiene especially in orthodontic patients.

Orthodontic patients face challenges with mechanical plaque removal, requiring various strategies to control plaque formation, prevent gingivitis, and maintain the periodontal health.8 Mechanical plaque removal with toothbrushes and interdental devices is the most common method for controlling plaque at home. Most patients prefer manual toothbrushes, whether conventional or orthodontic, due to their lower cost and ease of use. Although powered toothbrushes are more effective than manual ones in reducing plaque and gingivitis both short and long term in non-orthodontic patients, the effectiveness of powered versus manual toothbrushes is still uncertain for the orthodontic patients. A recent systematic review and meta-analysis concluded that there was no significant difference between manual and powered toothbrushes in reducing plaque accumulation or gingivitis in patients with fixed orthodontic devices.9 Selecting oral hygiene instruments that are most appropriate for each patient's specific needs is crucial for motivating orthodontic patients. Manual orthodontic toothbrushes have undergone advancements in bristle design and material. Many types of toothbrush options have been promoted for orthodontic patients. The use of orthodontic toothbrushes is currently preferred over other types of toothbrushes due to their bristle design, which makes it easier to clean the area around the brackets. Since orthodontic toothbrushes typically feature a V-shaped groove, while the shorter bristles within the groove are designed to clean the middle bracket area, the longer bristles are intended to clean the surroundings of the brackets. Studies comparing the effectiveness of orthodontic and conventional toothbrushes in reducing plaque and gingivitis on teeth with fixed appliances have shown conflicting results.8,10-12 More recently, single-tufted brushes have been investigated for their effectiveness in plaque removal. Single-tufted toothbrushes are recommended as an adjunctive device for surfaces and areas of the teeth that are not easily reached with other oral hygiene devices, such as the distal surfaces of molars, furcation areas, irregular gingival margins and areas of crowded teeth.13,14 Hasegawa et al., who first compared the effectiveness of single-tufted toothbrushes with the golden standard conventional toothbrush in controlling newly formed biofilm in the dentogingival area of healthy individuals, found it effective at controlling short-term dental biofilm neoformation on the dentogingival area.15 There are limited studies comparing the plaque removal efficacy of single-tufted brushes with conventional toothbrushes15,16, and one study has investigated in orthodontic patients.17 However, none of them has monitored their periodontal health in the long term and have compared single-tufted toothbrushes with conventional and orthodontic toothbrushes together. It was hypothesized that single-tufted toothbrushes are more effective in plaque removal and the healing of gingival inflammation than conventional toothbrushes and as effective as orthodontic toothbrushes. Therefore, it was aimed to evaluate the long-term effectiveness of different toothbrushes in removing plaque and gingival inflammation in individuals under fixed orthodontic treatment for gingivitis.

ELIGIBILITY:
Inclusion criteria:

* patients who had at least 22 teeth with brackets (excluding third molars)
* 18-35 yo
* had a diagnosis of dental plaque biofilm-induced gingivitis defined as ≥10% of --sites with bleeding on probing (BoP) and mean probing depth (PD) ≤3 mm
* were systemically healthy, non-smokers, or smoked <10 cigarettes per day for at least five years
* had not used antibiotics for the last three months
* were not pregnant.

Exclusion criteria:

* patients who smoked ≥ 10 cigarettes per day for at least five years
* who had less than 26 teeth with brackets
* were younger than 18 years of age or older than 35 years of age
* were periodontally healthy or had periodontitis
* who had systemic disease
* had used antibiotics in the last three months were pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Gingival inflammation | at the baseline, first week, sixth week and third month
  Löe & Silnesss Gingival index
bleeding on probing | at the baseline, first week, sixth week and third month
  bleeding on probing

SECONDARY OUTCOMES:
Dental biofilm | at the baseline, first week, sixth week and third month
  Turesky modification of Quigley-Hein plaque Index

OTHER OUTCOMES:
Pocket depth | at the baseline, first week, sixth week and third month
  Measuring probing pocket depth by a North Carolina periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University Dental Hospital, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The authors have not yet decided on data sharing. Revisions will be made when it is determined on which website it can be published.

REFERENCES:
- [Result] Lee DW, Moon IS. The plaque-removing efficacy of a single-tufted brush on the lingual and buccal surfaces of the molars. J Periodontal Implant Sci. 2011 Jun;41(3):131-4. doi: 10.5051/jpis.2011.41.3.131. Epub 2011 Jun 30. PMID 21811688
- [Result] Rafe Z, Vardimon A, Ashkenazi M. Comparative study of 3 types of toothbrushes in patients with fixed orthodontic appliances. Am J Orthod Dentofacial Orthop. 2006 Jul;130(1):92-5. doi: 10.1016/j.ajodo.2006.01.018. PMID 16849078
- [Result] ElShehaby M, Mofti B, Montasser MA, Bearn D. Powered vs manual tooth brushing in patients with fixed orthodontic appliances: A systematic review and meta-analysis. Am J Orthod Dentofacial Orthop. 2020 Nov;158(5):639-649. doi: 10.1016/j.ajodo.2020.04.018. Epub 2020 Sep 17. PMID 32951930
- [Result] Ericsson I, Thilander B, Lindhe J. Periodontal conditions after orthodontic tooth movements in the dog. Angle Orthod. 1978 Jul;48(3):210-8. doi: 10.1043/0003-3219(1978)0482.0.CO;2. No abstract available. PMID 280130
- [Result] Axelsson P, Nystrom B, Lindhe J. The long-term effect of a plaque control program on tooth mortality, caries and periodontal disease in adults. Results after 30 years of maintenance. J Clin Periodontol. 2004 Sep;31(9):749-57. doi: 10.1111/j.1600-051X.2004.00563.x. PMID 15312097
- [Result] Diamanti-Kipioti A, Gusberti FA, Lang NP. Clinical and microbiological effects of fixed orthodontic appliances. J Clin Periodontol. 1987 Jul;14(6):326-33. doi: 10.1111/j.1600-051x.1987.tb00979.x. PMID 3509967
- [Result] Zachrisson S, Zachrisson BU. Gingival condition associated with orthodontic treatment. Angle Orthod. 1972 Jan;42(1):26-34. doi: 10.1043/0003-3219(1972)0422.0.CO;2. No abstract available. PMID 4500561
- [Derived] Aykol-Sahin G, Ay-Kocabas B, Mert B, Usta H. Effectiveness of different types of toothbrushes on periodontal health in orthodontic patients with gingivitis: A randomized controlled study. BMC Oral Health. 2024 Oct 25;24(1):1289. doi: 10.1186/s12903-024-05084-x. PMID 39455996